CLINICAL TRIAL: NCT05867979
Title: Search for Structural Variants in Patients With Disorders of Sex Development (DSD) and Inconclusive Molecular Diagnosis GENEXPLOR-DSD
Brief Title: Search for Structural Variants in Patients With DSD and Inconclusive Molecular Diagnosis
Acronym: GENEXPLOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL22_0236; 2022-A02498-35 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2023-05-02; First posted 2023-05-22 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Disorder of Sex Development, 46,XY
MeSH Terms: conditions — Disorder of Sex Development, 46,XY

STUDY DESIGN:
Intervention Model Description: This is a single-center molecular biology pilot study on a single group of 20 patients with a disorder of sex development and inconclusive molecular diagnosis.
  The 20 blood samples from patients with severe or moderate DSD, with an inconclusive diagnosis will benefit from the Optical Genome Mapping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients with DSD and inconclusive molecular diagnosis (Experimental): The one arm of the study will have a venous blood draw as part of the research. 1 EDTA tube of 5mL will be collected.
  Interventions: Diagnostic Test: Identify structural variants by Optical Genome Mapping of DNA extracted from blood leukocytes

INTERVENTIONS:
Diagnostic Test: Identify structural variants by Optical Genome Mapping of DNA extracted from blood leukocytes — The one arm of the study will have a venous blood draw as part of the research. 1 EDTA tube of 5mL will be collected.

SUMMARY:
The goal of this clinical trial is to identify structural variants by Optical Genome Mapping (OGM) in the described participant population.

The main questions it aims to answer are:

* Identify constitutional structural variants by OGM of DNA extracted from blood leukocytes of patients with DSD for which the molecular diagnosis is inconclusive.
* Identify mosaic structural variants (present in a subpopulation of somatic cells only) by OGM of DNA extracted from blood leukocytes of patients with DSD for which the molecular diagnosis is inconclusive.
* Compare the diagnostic yields of OGM and of Comparative Genome Hybridization Array (CGH array) methods.
* Compare the diagnostic yields of the OGM and of Whole Genome Sequencing (National Sequencing Program), only if performed.

Participants will be required to:

* a follow-up interview with a physician to review their own and family medical and surgical history, with a focusing on DSD.
* An interview to assess their exposure to environmental pollutants during fetal life, using a validated questionnaire.
* a blood test with a 5mL tube to perform optical genome mapping analysis.

DETAILED DESCRIPTION:
Patients with severe or moderate disorder of sex development (DSD) with a inconclusive molecular diagnosis will benefit from optical genome mapping analysis.

A venous blood sample on ethylenediaminetetraacetic acid (EDTA) tube (5mL) will be taken in order to extract the DNA that will be used for the optical genome mapping analysis.

ELIGIBILITY:
Inclusion Criteria:

* homogeneous XY male karyotype.
* patient at least 6 months old
* severe to moderate DSD (Prader 1 to 5) for which the molecular diagnosis is inconclusive after a gene panel analysis.

Exclusion Criteria:

* subject with a homogeneous or mosaic XX, or monosomal X karyotype.
* subject with an aneuploidy.
* subject with a conclusive molecular diagnosis explaining the observed DSD (i.e. carrier of a causal genotype already well characterized by functional studies)

Min Age: 6 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — XY male karyotype (i.e. on all leukocytes studied).
Enrollment: 20 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a constitutional structural variants detected by OGM | Day of inclusion
  A structural variant, present at the constitutional state in leukocyte DNA, and considered as likely pathogenic or pathogenic, identified by OGM in at least one of the included patients.

SECONDARY OUTCOMES:
Number of Participants with mosaic structural variants detected by OGM | Day of inclusion
  A structural variant, present at the mosaic state in leukocyte DNA (i.e. allelic imbalance less than 0.40), and considered as likely pathogenic or pathogenic, identified by OGM in at least one of the included patients.

CONTACTS AND LOCATIONS:
Overall Officials: Françoise PARIS, MD PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No